CLINICAL TRIAL: NCT03122002
Title: A Prospective Cohort Study of Predictors and Prognostic Factors on the Acute Ischemic Stroke
Brief Title: Predictors and Prognostic Factors on the Acute Ischemic Stroke
Status: Terminated | Type: Observational
Why Stopped: Limited number of participants enrolled.
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wei Wang, Vice President of Tongji Hospital, Tongji Hospital
Other Study IDs: Know more about AIS
Record Dates: First submitted 2017-03-30; First posted 2017-04-20 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Cerebral Infarction; Cerebrovascular Disorders
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction; Cerebrovascular Disorders | interventions — Drug Therapy; Aspirin; Clopidogrel; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Emergency Treatment; Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients With Ischemic Stroke: The patients with all types of ischemic stroke including TIA, small vessle diseases, MCAO, and ect. These patients will be recorded their emergency treatment, medical history, details about their drug therapy, results of their routine blood test and image scan, and whether they receive intravascular therapy in time or not.
  Interventions: Drug: Drug Therapy; Diagnostic Test: Routine Blood Test and Image Scan; Other: Intravascular therapy; Other: Emergency Treatment; Other: Medical history
- Healthy Control: The patients admitted to hospital for symptoms like dizzness and headache, which later proved to be not related to cerebral vascular diseases, would be treated as control. Their medical history and the results of their routine blood test and image scan will be recorded.
  Interventions: Diagnostic Test: Routine Blood Test and Image Scan; Other: Medical history

INTERVENTIONS:
Drug: Drug Therapy — For this observation research, anti platelet drugs, statins and ect. would be used as clinical guidelines as usal, and statical ananysis of the relationship between these drugs and the final outcomes
  Other Names: Aspirin; Clopidogrel; Statin
  Groups: Patients With Ischemic Stroke
Diagnostic Test: Routine Blood Test and Image Scan — Routine blood test(HCY, LDL and ect.) and image scan (DWI, DSA and ect.)
Other: Intravascular therapy — Intravascular therapy including thrombectomy
  Groups: Patients With Ischemic Stroke
Other: Emergency Treatment — Emergency treatment including time to self-diagnosis of stroke, time to call for help, devices used to hospital and ect.
  Groups: Patients With Ischemic Stroke
Other: Medical history — Medical history including hypertension, diabetes, hyperlipemia and ect.

SUMMARY:
Through 5 years continuous observation of acute ischemic stroke patients in Neurology Department of Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, clinical data about emergency treatment (neurological score, examination and treatment), medical data after admission (neurological score, inspection, examination and treatment) and long-term prognosis (neurological score) was collected. The outcomes were set as the score scale, all blood test index and examination index of the research objects at specific period after illness. Through statistical analysis and comparison of different in-hospital clinical data in predicting the outcome of the patients, our study will provide more evidence-based solutions for the treatment and prediction of acute ischemic stroke.

DETAILED DESCRIPTION:
The research is designed as registrated, prospective, open-labeled, blind-endpoint, and the research objects are continuously recorded. The final subgroups are blind to neurological evaluators, data inputers and statisticians.

The research is a continuous observational exploratory study. All patients with ischemic stroke admitted to Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology from April 1, 2017 to December 31, 2021 will be included. According to the current situation, it is expected to enroll approximately 5000 of eligible patients for long-term follow-up observation.

We'll use multiple linear regression analysis model to study factors and confounding factors and their interaction. And we will control the confounding factors, and make a quantitative description of the relationship between factors and outcome variables.

Missing cases will be treated as censored values, and the ratio of missing cases will be recorded. All samples will be analyzed by Intent-to-Treat (ITT) analysis. In the analysis, if the results are statistically significant, the missing cases in the exposed group will be deleted, and the missing cases in non-exposure group be added. If the results are still statistically significant, then the missing cases are defined as not affecting the analysis results.

If the heterogeneity of data is large, the objects will be analyzed in subgroups according to age or sex.

If the missing rate is greater than 20%, it is necessary to analyze the sensitivity of the whole sample.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old, of either sex
* Confirmation by CT scan
* Willingness to participate in the study and comply with its procedures by signing a written informed consent

Exclusion Criteria:

* Cerebral hemorrhagic infarction confirmed by CT scan
* Patients with severe systemic disease who are expected to survive for no more than three months
* Unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ischemic stroke admitted to Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology from April 1, 2017 to December 31, 2021 will be included.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale scores | Change from Baseline mRS score at 24 months
  0 = No symptoms; 1 = No significant disability. Able to carry out all usual activities, despite some symptoms; 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 = Moderate disability. Requires some help, but able to walk unassisted; 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 = Dead.

SECONDARY OUTCOMES:
Re-admission to the hospital | 24 months
  Re-admission to the hospital (patients without new symptoms and admitted to the hospital simply for physical examination are not counted)
Cerebral and Cardio vascular diseases | 24 months
  Cerebral and Cardio vascular diseases including small vessel diseases, white matter ischemia, micro hemorrhage, ischemic stroke and hemorrhagic stroke.
Neurological deterioration-1 | Change from Baseline NIHSS score at 24 months
  Neurological deterioration (NIHSS score)
Neurological deterioration-2 | Change from Baseline FAQ score at 24 months
  Neurological deterioration (FAQ score)
Cognitive dysfunction | Change from Baseline MMSE score at 24 months
  Cognitive dysfunction (MMSE score). Patients with cognitive dysfunction will be classified into mild neurocognitive disorder, major neurocognitive disorder according to DSM-5
Cognitive dysfunction | Change from Baseline MoCA score at 24 months
  Cognitive dysfunction (MoCA score). Patients with cognitive dysfunction will be classified into mild neurocognitive disorder, major neurocognitive disorder according to DSM-5
Cerebrospinal Fluid (CSF) test | 24 months
  Cerebrospinal Fluid (CSF) test including Tau, Aβ and ect.
Blood test | 24 months
  Blood including HCY, amino acid, LDL and ect.
Depression | 24 months
  Hamilton Depression Scale
Severe pulmonary infection | 24 months
  Severe pulmonary infection

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, PhD, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shang K, Chen X, Cheng C, Luo X, Xu S, Wang W, Liu C. Arterial Tortuosity and Its Correlation with White Matter Hyperintensities in Acute Ischemic Stroke. Neural Plast. 2022 Mar 24;2022:4280410. doi: 10.1155/2022/4280410. eCollection 2022. PMID 35369646
- [Derived] Qin C, Zhao XL, Ma XT, Zhou LQ, Wu LJ, Shang K, Wang W, Tian DS. Proteomic profiling of plasma biomarkers in acute ischemic stroke due to large vessel occlusion. J Transl Med. 2019 Jul 1;17(1):214. doi: 10.1186/s12967-019-1962-8. PMID 31262327